CLINICAL TRIAL: NCT07144059
Title: Participants Are Not Assigned to Interventions Based on a Protocol
Brief Title: Impact of Non-medicalized ECG Practices Initiated by SAMU in Dispatch Strategies
Acronym: ECG-PHNM
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0017
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute coronary syndrome; infarct; STEMI; Electrocardiogram (ECG); Coronary angiography; SAMU; SMUR; Non-medical vectors
MeSH Terms: conditions — Acute Coronary Syndrome; Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EMS Vector: Patients who had the qualifying ECG by the SMUR after medical interrogation by the SAMU
  Interventions: Other: ECG by the SMUR after medical interrogation by the SAMU
- ECG Vector: SP/Ambulances: Patients who have called the emergency services with either an ECG performed by a non-medical vector (SP or ambulance), or a decision to reinforce SMUR during the first aid assessment
  Interventions: Other: ECG performed by a non-medical vector

INTERVENTIONS:
Other: ECG by the SMUR after medical interrogation by the SAMU — Patients who had the qualifying ECG by the SMUR after medical interrogation by the SAMU
  Groups: EMS Vector
Other: ECG performed by a non-medical vector — Patients who have called the emergency services with either an ECG performed by a non-medical vector (SP or ambulance), or a decision to reinforce SMUR during the first aid assessment
  Groups: ECG Vector: SP/Ambulances

SUMMARY:
The performance of an ECG by non-medicalized prehospital teams (firefighters, first responders, paramedic ambulances) is developing across the territory to cope with the increasing demand (SAMU calls) for a service that cannot meet it (limited Mobile Emergency and Resuscitation Unit - SMUR - teams).

Early diagnosis of acute coronary syndrome is key to appropriate management. A delay in care can quickly lead to complications ranging from rhythm disorders to cardiac arrest. Furthermore, as with reperfusion in strokes, the earlier reperfusion treatment is initiated, the greater the beneficial effect in ST-segment elevation myocardial infarction (STEMI).

Moreover, the main elements for diagnosing STEMI in the prehospital setting remain the ECG, along with the anamnesis (medical history) and clinical examination (typical pain).

This is an observational, retrospective and single-center study (SAMU 91) carried out between September 1, 2023 and December 31, 2024. The inclusion criteria for our study were adult patients who had been regulated by SAMU 91 during a primary intervention and who had ST+ ACS registered in the eMUST registry. The main objective was to study the difference in the admission times of patients admitted to the emergency intensive care unit of cardiology or coronary angiography and presenting with ST+ ACS on the ECG performed by a primary SMUR team versus a non-medical team referred by the SAMU. The secondary objectives were to study the descriptive variables between the two groups (SMUR and non-medicalized vector), the typicity of pain, the mortality rate and the morbidity rate between the two groups.

DETAILED DESCRIPTION:
The list of patients with ST+ ACS in department 91 during the year 2023 and 2024 were extracted from the E-Must registry (Registry for the Evaluation in Emergency Medicine of Therapeutic Strategies for Myocardial Infarction of less than 24 hours treated by the SAMU/SMUR of Île-de-France) and the missing information was retrieved via the SAMUScript medical regulation software (call schedules, address of the place of intervention,...)

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient regulated by the SAMU 91 between 09/2023 and 12/2024
* Patient referred for coronary angiography for ST+ ACS
* Patient registered in the E-Must register (Registry for the Evaluation in Emergency Medicine of Therapeutic Strategies for Myocardial Infarction of less than 24 hours treated by the SAMU/SMUR of Île-de-France)

Exclusion Criteria:

* Secondary transport

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients regulated by the SAMU 91 in primary intervention in the Essonne department with ST+ ACS and admitted to the ICU or coronary angiography department
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Coronary Angiography or Cardiology Intensive Care Admission | day 0
  Time between the time of the call for help and the arrival in the coronary angiography department or cardiology intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Patrick HU, MD, Study Director — Centre Hospitalier Sud Francilien

IPD SHARING:
Plan to Share IPD: No